CLINICAL TRIAL: NCT03365466
Title: Anticoagulation Therapies Effect on the Endometrial Blood Flow and Pregnancy Outcomes in Unexplained Recurrent Implantation Failure Women
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Principal Investigator, Shihua Bao, Principal Investigator, Shanghai First Maternity and Infant Hospital
Other Study IDs: ShanghaiFMIH-uRIF
Record Dates: First submitted 2017-12-02; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-09

CONDITIONS: Recurrent Implantation Failure
Keywords: recurrent implantation failure; aspirin; low molecular weight heparin
MeSH Terms: interventions — Aspirin; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group A: Patients who received a daily dose of 75mg LDA per day after menstruation prior to ET.
  Interventions: Drug: Low dose aspirin
- Group B: Patients who received a daily dose of 5000u LMWH after menstruation prior to ET.
  Interventions: Drug: Low molecular weight heparin
- Group C: Patients who received a daily dose of 75 mg LDA plus 5000u LMWH after menstruation prior to ET.
  Interventions: Drug: Low dose aspirin plus low molecular weight heparin
- Group D: Patients who did not receive any treatment.
  Interventions: Drug: no treatment

INTERVENTIONS:
Drug: Low dose aspirin — LDA 25mg tid
  Groups: Group A
Drug: Low molecular weight heparin — LMWH 5000u IH qd
  Groups: Group B
Drug: Low dose aspirin plus low molecular weight heparin — LDA 25mg tid + LMWH 5000u IH qd
  Groups: Group C
Drug: no treatment — Patients who did not receive any treatment.
  Groups: Group D

SUMMARY:
The aim of the study is to investigate whether Low Dose Aspirin and Low Molecular Weight Heparin could increase the uterine perfusion, and finally improve the implantation and pregnancy rates in patients with unexplained recurrent implantation failure.

DETAILED DESCRIPTION:
Infertility is a growing issue for many couples all over the world. Nowadays, Assisted reproductive technology is widely used to treat couples affected by infertility, but, the success rate is still very low. Recurrent implantation failure is an important cause of repeated IVF failure. In addition to the embryo quality, a functioning and receptive endometrium is crucial for embryo implantation. There is a growing amount of evidence shows that uterine perfusion playing an important part in regulating endometrial receptivity and in successful pregnancy.

Recently, transvaginal ultrasonography is often used to examine endometrial thickness, pattern and blood flow status to predict uterine receptivity. Some studies have demonstrated that uterine artery blood flow resistance in RM (Recurrent miscarriage) patients is significantly higher than in normal fertile patients. It has been postulated that abnormal uterine perfusion could be related to the reproductive failure, enhancing the uterine perfusion may improve the successful pregnancy. In accordance with this hypothesis, some therapeutic approaches including low dose aspirin (LDA), nitric oxide donor, low molecular weight heparin, sildenafil are applying in clinic. Low molecular weight heparin (LMWH) is derived from unfractionated heparin. It also has anticoagulation or the antithrombin effect. Aspirin has analgesic, antipyretic, and anti-inflammatory properties. Initially, aspirin and low molecular weight heparin have been used either as single agents or in combination to treat patients with recurrent miscarriage, diagnosed with antiphospholipid syndrome. The treatment confers a significant benefit in live births rate. Furthermore, various studies have shown that thrombophilia are more common in women with RIF compared with healthy fertile controls. In these women, heparin treatment could potentially enhance the implantation process, and may finally improve the live birth rate. The aim of the study is to investigate whether Low Dose Aspirin and Low Molecular Weight Heparin could increase the uterine perfusion, and finally improve the implantation and pregnancy rates in patients with unexplained recurrent implantation failure.

ELIGIBILITY:
Inclusion Criteria:

1. ≥3 pervious IVF-ET failures or failure with transfer of at least 10 frozen embryos in multiple transfers;
2. 25-45 years old;
3. Having a regular menstrual cycle and BBT;
4. Top-quality frozen embryos for transfer;
5. Endometrial thickness 8-14mm；
6. Abnormal uterine perfusion(PI>2.5)；
7. Decided to recieve LMWH or LDA or a combination of LMWH and LDA therapy.

Exclusion Criteria:

1. Chromosome aberrations in anyone of the couple;
2. Abnormal uterine cavity;
3. Hydrosalpinx;
4. Chronic systemic disease(liver,renal,heart,thyroid and thrombocytopenia)
5. Having experienced severe allergies, trauma history；
6. With a history of mental illness;
7. Any contraindication for LDA or LMWH.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This is a prospective cohort study on unexplained recurrent implantation failure patients with abnormal uterine perfusion in our clinic from September 2017 to December 2018.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | until 12 weeks
  Ongoing pregnancy beyond the 12th gestational week rate

SECONDARY OUTCOMES:
Uterine artery blood flow | luteal phase before ET and one day before ET
  by transvaginal sonography
Implantation rate | 8 weeks
  by transvaginal sonography

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai first Maternity and Infant health hospital, Tong Ji University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No